CLINICAL TRIAL: NCT00175253
Title: Alemtuzumab Induction With Tacrolimus and MMF Maintenance Immunosuppression in Islet Transplantation
Brief Title: Alemtuzumab Induction in Islet Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5369
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Type 1 Diabetes
Keywords: islet; transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Alemtuzumab

INTERVENTIONS:
Drug: alemtuzumab
Procedure: islet transplant

SUMMARY:
Our experience suggests that further research with alemtuzumab is attractive in islet transplantation. Therefore, in this study we propose to combine alemtuzumab induction pre-transplant, with tacrolimus and mycophenolate mofetil maintenance immunosuppression post-transplant. In the critical early phase post transplant, we anticipate that this regimen will prove to be more effective in control of autoimmunity or rejection events, and have a more desirable side-effect profile, than previously tested combinations of induction and immunosuppressive agents.

DETAILED DESCRIPTION:
This trial is a single-center, prospective, open-label study in 12 Type 1 diabetic participants receiving an islet-alone transplant along with alemtuzumab induction therapy followed by combination tacrolimus and MMF maintenance immunosuppression. Participants will receive 1 to 3 infusions of pancreatic islets of sufficient quantity to attain insulin independence.

The primary objective of this protocol is to assess the safety of a treatment regimen utilizing alemtuzumab induction and a combination of tacrolimus and MMF maintenance immunosuppression in adult Type 1 diabetic participants receiving their first islet transplant.

ELIGIBILITY:
Inclusion Criteria:

* open to Canadians only
* participant must have had Type 1 diabetes mellitus for more than 5 years
* diabetes must be complicated by at least 1 of the following situations that persist despite intensive insulin management efforts: (1) Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 2 or more episodes of severe hypoglycemia requiring third party assistance within 12 months; or (2) Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 2 or more hospital visits for diabetic ketoacidosis over the last 12 months.
* Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* Severe co-existing cardiac disease
* Active alcohol or substance abuse, to include cigarette smoking
* Psychiatric disorder making the subject not a suitable candidate for transplantation
* History of non-adherence to prescribed regimens
* Active infection including Hepatitis C, Hepatitis B, HIV, TB
* Any history of or current malignancies except squamous or basal skin cancer
* BMI > 28 kg/m2 at screening visit
* Creatinine clearance < 65 mL/min/1.73 m2
* Blood creatinine > 150 µmol/L (1.7 mg/dL)
* Macroalbuminuria (urinary albumin excretion rate > 300 mg/24h)
* Baseline Hb < 105g/L (<10.5 g/dL) in women, or < 130 g/L (<13 g/dL) in men
* Baseline screening liver function tests outside of normal range
* Untreated proliferative retinopathy
* Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast feeding
* Previous transplant, or evidence of significant sensitization on PRA
* Insulin requirement >1.0 U/kg/day
* HbA1C >12%
* Uncontrolled hyperlipidemia
* Under treatment for a medical condition requiring chronic use of steroids
* Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT INR > 1.5
* Untreated Celiac disease
* Patients with Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-11; Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A.M. James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta - Clinical Islet Transplant Program, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Gala-Lopez B, Kin T, O'Gorman D, Pepper AR, Senior P, Humar A, Shapiro AM. Microbial contamination of clinical islet transplant preparations is associated with very low risk of infection. Diabetes Technol Ther. 2013 Apr;15(4):323-7. doi: 10.1089/dia.2012.0297. Epub 2013 Feb 25. PMID 23438305